CLINICAL TRIAL: NCT02468986
Title: Analysis of Endothelial Cells in Rheumatoid Arthritis
Brief Title: Study of Venous Endothelial Cells in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Elizabeth Blair Solow, ASSISTANT PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU 012011-034
Record Dates: First submitted 2014-03-06; First posted 2015-06-11 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum collected by serum separator tube. Will be processed and frozen at -80degrees.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Uncontrolled Rheumatoid Arthritis: 18-75 years old; Rheumatoid arthritis, defined by 1987 American College Rheumatology criteria; Attending clinic at Aston Center for Rheumatology or Parkland Rheumatology Clinic; Uncontrolled: Patients will be labeled as uncontrolled RA if Disease Activity Score (DAS) score is >3.2 and C-reactive protein (mg/dL) elevated above normal range.
  Excluding: Insulin dependent diabetes; Cardiovascular or Cerebrovascular disease (history of myocardial infarction, stroke, peripheral vascular disease); Tobacco use in the past 24 months; Uncontrolled hypertension (BP > 150/90) in the past 3 months; Uncontrolled hyperlipidemia (LDL>160) in the past 6 months; Pregnant or nursing.
- Controlled Rheumatoid Arthritis: 18-75 years old; Rheumatoid arthritis, defined by 1987 American College Rheumatology criteria; Attending clinic at Aston Center for Rheumatology or Parkland Rheumatology Clinic; Controlled: Disease activity score (DAS) <3.2, normal C-reactive protein. Excluding: Insulin dependent diabetes; Cardiovascular or Cerebrovascular disease (history of myocardial infarction, stroke, peripheral vascular disease); Tobacco use in the past 24 months; Uncontrolled hypertension (BP > 150/90) in the past 3 months; Uncontrolled hyperlipidemia (LDL>160) in the past 6 months; Pregnant or nursing.
- Healthy Controls: 18-75 years old. Excluding: Insulin dependent diabetes; Cardiovascular or Cerebrovascular disease (history of myocardial infarction, stroke, peripheral vascular disease); Tobacco use in the past 24 months; Uncontrolled hypertension (BP > 150/90) in the past 3 months; Uncontrolled hyperlipidemia (LDL>160) in the past 6 months; Pregnant or nursing.

SUMMARY:
Heart disease is the major contributor of early death in rheumatoid arthritis (RA) and is not influenced by traditional risk factors. Blood vessel dysfunction has been associated with heart disease and complications such as heart attack. The vessel dysfunction is thought to be mediated in part to inflammation. RA patients have evidence of vessel dysfunction seen on ultrasound that improves after medications are given.

The purpose of this study is to evaluate patients with controlled or uncontrolled rheumatoid arthritis to determine if there is a difference in the protein expression in the cells that line the blood vessels compared to healthy people.

DETAILED DESCRIPTION:
The study will consist of a cross sectional analysis of venous endothelial cells in rheumatoid arthritis patients who have controlled or uncontrolled disease and healthy controls. We will collect venous endothelial cells by placing an IV in antegrade position in the forearm and a thin wire will be inserted to collect the cells from the inner lining of the vein. The cells will processed and stained for markers of endothelial function and oxidative stress including endothelial nitric oxide synthase (eNOS), phospho-eNOS, nuclear factor kappa B (NFκB), and nitrotyrosine using immunofluorescence technique. Flow mediated dilation (FMD) by ultrasound of the brachial artery on the contralateral arm will be used as an additional marker of endothelial function. A blood sample will be taken for analysis of inflammatory markers (sedimentation rate, C-reactive protein) and cytokine analysis (IL-1, IL-6, TNFa) by cytokine bead array and flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

Rheumatoid arthritis:

* Age 18-75 years
* Rheumatoid arthritis defined by 1987 American College of Rheumatology criteria
* Attending clinic at University of Texas Southwestern Aston Clinic for Rheumatology or Parkland Arthritis Clinic.

Healthy controls:

- Age 18-75 years.

Exclusion Criteria:

Rheumatoid arthritis:

* Insulin dependent diabetes
* Cardiovascular or Cerebrovascular disease
* Tobacco use in last 24 months
* Uncontrolled blood pressure
* Uncontrolled cholesterol
* Pregnant or nursing
* Prednisone greater than 10mg per day
* Stable methotrexate dose for less than 4 weeks
* Undergoing Infliximab infusions

Healthy controls:

* Insulin dependent diabetes
* Cardiovascular or Cerebrovascular disease
* Tobacco use in last 24 months
* Uncontrolled high blood pressure
* Uncontrolled cholesterol
* Pregnant or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients will be selected from arthritis clinics associated with UT Southwestern Medical Center and Parkland Memorial Hospital. Healthy controls will be collected from primary care clinics who refer to these specialty clinics.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Endothelial cell protein expression by immunofluorescence microscopy of endothelial nitric oxide synthase, nitrotyrosine, nuclear factor kappa B. | Cells are immediately processed following extraction and placed in -80 degree C freezer. Cells are then analyzed by immunofluorescence microscopy in batches of subjects. Patient is followed-up 24 hours after by phone.
  Immunofluorescence microscopy of frozen endothelial cells will be processed in batches to reduce bias. Cells are assessed for individual protein expression at study entry. Repeated collection of cells will not been done.

SECONDARY OUTCOMES:
Serum cytokines analysis by cytometric bead array | Measured once upon enrollment into study. Patient is followed-up 24 hours after by phone.
  Interleukin-1, Interleukin-6, Tumor Necrosis Factor -alpha
Flow mediated dilation assessed in the brachial artery by ultrasound | Measured once upon enrollment into study. Patient is followed-up 24 hours after by phone.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Solow, MD, Principal Investigator — University of Texas; David Karp, MD, PhD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas

REFERENCES:
- [Background] Vaudo G, Marchesi S, Gerli R, Allegrucci R, Giordano A, Siepi D, Pirro M, Shoenfeld Y, Schillaci G, Mannarino E. Endothelial dysfunction in young patients with rheumatoid arthritis and low disease activity. Ann Rheum Dis. 2004 Jan;63(1):31-5. doi: 10.1136/ard.2003.007740. PMID 14672888
- [Background] Maradit-Kremers H, Crowson CS, Nicola PJ, Ballman KV, Roger VL, Jacobsen SJ, Gabriel SE. Increased unrecognized coronary heart disease and sudden deaths in rheumatoid arthritis: a population-based cohort study. Arthritis Rheum. 2005 Feb;52(2):402-11. doi: 10.1002/art.20853. PMID 15693010
- [Background] del Rincon ID, Williams K, Stern MP, Freeman GL, Escalante A. High incidence of cardiovascular events in a rheumatoid arthritis cohort not explained by traditional cardiac risk factors. Arthritis Rheum. 2001 Dec;44(12):2737-45. doi: 10.1002/1529-0131(200112)44:123.0.CO;2-%23. PMID 11762933
- [Background] Neunteufl T, Katzenschlager R, Hassan A, Klaar U, Schwarzacher S, Glogar D, Bauer P, Weidinger F. Systemic endothelial dysfunction is related to the extent and severity of coronary artery disease. Atherosclerosis. 1997 Feb 28;129(1):111-8. doi: 10.1016/s0021-9150(96)06018-2. PMID 9069525
- [Background] Gonzalez-Juanatey C, Llorca J, Sanchez-Andrade A, Garcia-Porrua C, Martin J, Gonzalez-Gay MA. Short-term adalimumab therapy improves endo-thelial function in patients with rheumatoid arthritis refractory to infliximab. Clin Exp Rheumatol. 2006 May-Jun;24(3):309-12. PMID 16870100
- [Background] Galarraga B, Khan F, Kumar P, Pullar T, Belch JJ. C-reactive protein: the underlying cause of microvascular dysfunction in rheumatoid arthritis. Rheumatology (Oxford). 2008 Dec;47(12):1780-4. doi: 10.1093/rheumatology/ken386. Epub 2008 Oct 14. PMID 18854346
- [Background] Schwartz R, Osborne-Lawrence S, Hahner L, Gibson LL, Gormley AK, Vongpatanasin W, Zhu W, Word RA, Seetharam D, Black S, Samols D, Mineo C, Shaul PW. C-reactive protein downregulates endothelial NO synthase and attenuates reendothelialization in vivo in mice. Circ Res. 2007 May 25;100(10):1452-9. doi: 10.1161/01.RES.0000267745.03488.47. Epub 2007 Apr 19. PMID 17446434
- [Background] Oemar BS, Tschudi MR, Godoy N, Brovkovich V, Malinski T, Luscher TF. Reduced endothelial nitric oxide synthase expression and production in human atherosclerosis. Circulation. 1998 Jun 30;97(25):2494-8. doi: 10.1161/01.cir.97.25.2494. PMID 9657467